CLINICAL TRIAL: NCT04991844
Title: Healthy Eating for Successful Living in Older Adults™ Community Education Program
Brief Title: Healthy Eating for Successful Living in Older Adults Program (HE) Study
Acronym: HES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health and Healing Research Education and Service, Inc. (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 120180167
Record Dates: First submitted 2021-07-02; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Chronic Diseases, Multiple
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group did not receive any intervention, but met at three timepoints to complete study questionnaires and provide anthropometric measurements,
- Intervention Group (Experimental): This group received the study intervention protocol.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — Intervention group participants met once a week, for 2.5 hours, over a period of six weeks for the HES workshops. The HES workshops followed a scripted curriculum that incorporated information from the USDA's MyPlateTM, and the USDA 2015-2020 dietary guidelines. Participants were also taught goal-setting, problem-solving through brainstorming, group support, self-assessment and management of dietary and physical activity patterns.
  Arms: Intervention Group

SUMMARY:
The Healthy Eating for Successful Living in Older Adults™ (HESL) is a six-week community nutrition and lifestyle education program designed specifically for the elderly (>60 years), to promote dietary and behavioral changes towards a healthy lifestyle. The intervention was evaluated using a randomized-controlled trial.

DETAILED DESCRIPTION:
The elderly are at a higher risk of various chronic diseases. The burden of various chronic diseases such as heart disease and osteoporosis can be reduced with change in dietary and other lifestyle behaviors. The Healthy Eating for Successful Living in Older Adults™ (HESL) provides elderly with needed knowledge on healthy food choices and lifestyle behaviors, and tools that support behavioral changes. The investigators aimed to evaluate this intervention program by determining, among others, the impact of the intervention on factors such as dietary intake of fiber, and other nutrients, as well as healthy behaviors and food choices, and quality of life at 6 months post-intervention, using a randomized-controlled trial. The intervention group was compared to the control group receiving no intervention to evaluate the effects of the six-week HESL intervention on our outcome measures of interest.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate and complete all study activities following randomization into the intervention or control group.
* English-speaking.
* interested and able to participate.

Exclusion Criteria:

* None

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline dietary fiber intake at 6 months | 6 months post-intervention
  Change from baseline dietary fiber intake (mean intake in g/day) at 6 months using the Willett FFQ

SECONDARY OUTCOMES:
Change from baseline saturated fat intake at 6 months | 6 months post-intervention
  Change from baseline dietary saturated fat intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline polyunsaturated fat intake at 6 months | 6 months post-intervention
  Change from baseline dietary polyunsaturated fat intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline monounsaturated fat intake at 6 months | 6 months post-intervention
  Change from baseline dietary monounsaturated fat intake (mean intake in g/day) at 6 months using the Willett FFQ.
Change from baseline trans fat intake at 6 months | 6 months post-intervention
  Change from baseline dietary trans fat intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline cholesterol intake at 6 months | 6 months post-intervention
  Change from baseline dietary cholesterol intake (mean intake in mg/day) at 6 months using the Willett FFQ
Change from baseline omega-3 fat intake at 6 months | 6 months post-intervention
  Change from baseline dietary omega-3 fat intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline omega-6 fat intake at 6 months | 6 months post-intervention
  Change from baseline dietary omega-6 fat intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline calcium intake at 6 months | 6 months post-intervention
  Change from baseline dietary calcium intake (mean intake in mg/day) at 6 months using the Willett FFQ
Change from baseline vitamin D intake at 6 months | 6 months post-intervention
  Change from baseline dietary vitamin D intake (mean intake in IU/day) at 6 months using the Willett FFQ
Change from baseline folate intake at 6 months | 6 months post-intervention
  Change from baseline folate intake (mean intake in mcg/day) at 6 months using the Willett FFQ
Change from baseline potassium intake at 6 months | 6 months post-intervention
  Change from baseline potassium intake (mean intake in mg/day) at 6 months using the Willett FFQ
Change from baseline magnesium intake at 6 months | 6 months post-intervention
  Change from baseline magnesium intake (mean intake in mg/day) at 6 months using the Willett FFQ
Change from baseline vitamin B6 intake at 6 months | 6 months post-intervention
  Change from baseline vitamin B6 intake (mean intake in mg/day) at 6 months using the Willett FFQ
Change from baseline vitamin B12 intake at 6 months | 6 months post-intervention
  Change from baseline vitamin B12 intake (mean intake in mcg/day) at 6 months using the Willett FFQ
Change from baseline fruit intake at 6 months | 6 months post-intervention
  Change from baseline fruit intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline vegetable intake at 6 months | 6 months post-intervention
  Change from baseline vegetable intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline legume intake at 6 months | 6 months post-intervention
  Change from baseline legume intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline whole grain intake at 6 months | 6 months post-intervention
  Change from baseline whole grain intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline nut and seed intake at 6 months | 6 months post-intervention
  Change from baseline nut and seed intake (mean intake in g/day) at 6 months using the Willett FFQ
Change from baseline physical activity at 6 months | 6 months post-intervention
  Change from baseline physical activity (metabolic equivalent task (MET)-hours per week ) at 6 months using the Harvard Physical Activity Questionnaire.
Change from baseline Body mass index at 6 months (BMI, Kg/m2) | 6 months post-intervention
  Change from baseline Body mass index (calculated from: weight in kilograms, and height in meters; weight and height will be combined to report BMI, Kg/m2) at 6 months
Change from baseline quality of life measure at 6 months | 6 months post-intervention
  Change from baseline quality of life measure at 6 months using the Euro-QoL-5D-5L questionnaire; Participants were asked to provide a rating of their own health on a scale of 0-100, where 0 means "death" and 100 means "the best health.
Change in response to the question: "do you make food choices that are healthy for your bones?" from baseline at 6 months | 6 months post-intervention
  Change in response (in percentage points) to the above question at 6 months; questions were originally in a Likert scale from always to never with five categories. We converted responses into dummy variables (with 1=always, most of the time, or sometimes; and 0 =rarely and never).
Change in response to the question: "do you make food choices that are healthy for your heart?" from baseline at 6 months | 6 months post-intervention
  Change in response (in percentage points) to the above question at 6 months; questions were originally in a Likert scale from always to never with five categories. We converted responses into dummy variables (with 1=always, most of the time, or sometimes; and 0 =rarely and never).
Change in response to the question: "do you read nutrition labels when shopping or planning for meals?" from baseline at 6 months | 6 months post-intervention
  Change in response (in percentage points) to the above question at 6 months; questions were originally in a Likert scale from always to never with five categories. We converted responses into dummy variables (with 1=always, most of the time, or sometimes; and 0 =rarely and never).
Change in response to the question:"do you use MyPlateTM tools to help make food choices?" from baseline at 6 months | 6 months post-intervention
  Change in response (in percentage points) to the above question at 6 months; questions were originally in a Likert scale from always to never with five categories. We converted responses into dummy variables (with 1=always, most of the time, or sometimes; and 0 =rarely and never).
Change in response to the question: "How confident are you that you can manage most of your health problems?" from baseline at 6 months | 6 months post-intervention
  Change in response (in percentage points) to the above question at 6 months; questions were originally on a scale of 0-10, with 10 being most confident. These ratings were coded as 1 if they were 6 and above, and 0 if 5 or below.
Change in response to the question: "How understandable and useful is the information that your doctor or nurses have given you about your health problems or concerns?" from baseline at 6 months | 6 months post-intervention
  Change in response (in percentage points) to the above question at 6 months; questions were originally on a scale of 0-10, with 10 being most understandable/useful. These ratings were coded as 1 if they were 6 and above, and 0 if 5 or below.
Change in response to the sentence: "I play an active role in my health care and well-being." | 6 months post-intervention
  Change in response (in percentage points) to the above question at 6 months; questions were originally on a scale of 0-10, with 10 being most active. These ratings were coded as 1 if they were 6 and above, and 0 if 5 or below.

CONTACTS AND LOCATIONS:
Overall Officials: Junaidah Barnett, PhD, MCH(N), Principal Investigator — Health and Healing Research Education and Service, Inc.
Locations (1):
- Health and Healing Research Education and Service, Inc., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no such plans.

REFERENCES:
- [Derived] Barnett JB, Zeng W. Healthy Eating for Successful Living in Older Adults community education program-evaluation of lifestyle behaviors: A randomized controlled trial. Front Aging. 2022 Sep 6;3:960986. doi: 10.3389/fragi.2022.960986. eCollection 2022. PMID 36187849